CLINICAL TRIAL: NCT02931539
Title: A Phase 3, Multicenter, Randomized, Open-label, Active-controlled Study to Assess the Efficacy and Safety of Maribavir Treatment Compared to Investigator-assigned Treatment in Transplant Recipients With Cytomegalovirus (CMV) Infections That Are Refractory or Resistant to Treatment With Ganciclovir, Valganciclovir, Foscarnet, or Cidofovir
Brief Title: Efficacy and Safety Study of Maribavir Treatment Compared to Investigator-assigned Treatment in Transplant Recipients With Cytomegalovirus (CMV) Infections That Are Refractory or Resistant to Treatment With Ganciclovir, Valganciclovir, Foscarnet, or Cidofovir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP620-303; 2015-004725-13 (EudraCT Number)
Record Dates: First submitted 2016-09-29; First posted 2016-10-13 (Estimated); Results first posted 2021-09-23 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Cytomegalovirus (CMV)
MeSH Terms: interventions — maribavir; Ganciclovir; Valganciclovir; Foscarnet; Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maribavir Treatment (Experimental): Participants will receive 400 milligrams (mg) (2x200 mg tablets) maribavir twice daily orally (doses separated by a minimum of 8 hours) for 8 weeks.
  Interventions: Drug: Maribavir
- Investigator-Assigned Treatment (Active Comparator): Participants will receive anti-CMV agent best suited to treat the respective participant as per the investigator's prescribed dosing regimen for 8 weeks. Agents of choice include: ganciclovir, valganciclovir, foscarnet, or cidofovir.
  Interventions: Drug: Ganciclovir; Drug: Valganciclovir; Drug: Foscarnet; Drug: Cidofovir

INTERVENTIONS:
Drug: Maribavir — Maribavir 400 milligrams (mg) (2x200 mg tablets) will be administered twice daily for 8 weeks.
  Other Names: SHP620
  Arms: Maribavir Treatment
Drug: Ganciclovir — Ganciclovir as per the investigator's prescribed dosing regimen will be administered for 8 weeks.
  Arms: Investigator-Assigned Treatment
Drug: Valganciclovir — Valganciclovir as per the investigator's prescribed dosing regimen will be administered for 8 weeks.
  Arms: Investigator-Assigned Treatment
Drug: Foscarnet — Foscarnet as per the investigator's prescribed dosing regimen will be administered for 8 weeks.
  Arms: Investigator-Assigned Treatment
Drug: Cidofovir — Cidofovir as per the investigator's prescribed dosing regimen will be administered for 8 weeks.
  Arms: Investigator-Assigned Treatment

SUMMARY:
The purpose of this study is to compare the efficacy of maribavir to investigator-assigned anti-Cytomegalovirus (CMV) therapy in CMV viremia clearance in transplant recipients who are refractory or resistant to prior anti-CMV treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be able to provide written, personally signed, and dated informed consent to participate in the study before completing any study-related procedures. As applicable, a parent/both parents or legally authorized representative (LAR) must provide signature of informed consent and there must be documentation of assent by the participant before completing any study-related procedures.
2. The participant must be a recipient of hematopoietic stem cell or solid organ transplant.
3. The participant must have a documented CMV infection in whole blood or plasma, with a screening value of greater than or equal to (>=) 2730 international units per milliliter (IU/mL) in whole blood or >= 910 IU/mL in plasma in 2 consecutive assessments, separated by at least 1 day, as determined by local or central specialty laboratory quantitative polymerase chain reaction (qPCR) or comparable quantitative CMV DNA results. Both samples should be taken within 14 days prior to randomization with second sample obtained within 5 days prior to randomization. The same laboratory and same sample type (whole blood or plasma) must be used for these assessments.
4. The participant must have a current CMV infection that is refractory to the most recently administered of the four anti-CMV treatment agents. Refractory is defined as documented failure to achieve greater than (>) 1 log10 (common logarithm to base 10) decrease in CMV DNA level in whole blood or plasma after a 14 day or longer treatment period with intravenous (IV) ganciclovir/oral valganciclovir, IV foscarnet, or IV cidofovir.

   a. Participants with documentation of 1 or more CMV genetic mutations associated with resistance to ganciclovir/valganciclovir, foscarnet, and/or cidofovir must also meet the definition of refractory CMV infection.
5. The Investigator must be willing to treat the participant with at least one of the available anti-CMV drugs (ganciclovir, valganciclovir, foscarnet, or cidofovir). Note: Combination therapy with foscarnet and cidofovir is not permitted in the investigator-assigned anti-CMV treatment (IAT) arm due to the potential for serious nephrotoxicity.
6. The participant must be >= 12 years of age at the time of consent.
7. The participant must weigh >= 35 kilogram (kg).
8. The participant must have all of the following results as part of screening laboratory assessments (results from either the central laboratory or a local laboratory can be used for qualification):

   1. Absolute neutrophil count (ANC) >= 1000/ millimeter cube (mm^3) (1.0 x 10^9/liter [L])
   2. Platelet count >= 25,000/mm^3 [25 x 10^9/L],
   3. Hemoglobin >= 8 grams per deciliter (g/dL).
   4. Estimated glomerular filtration rate (eGFR) > 30 (milliliters per minute (mL/min) /1.73 square meter (m^2) as assessed by Modification of Diet in Renal Disease (MDRD) formula for participants >= 18 years of age or Schwartz formula for participants less than (<) 18 years of age.
9. The participant must have a negative serum beta-human chorionic gonadotropin (beta-HCG) pregnancy test at screening, if a female of child bearing potential. Additional urine pregnancy tests may be done per institutional requirements. Sexually active females of child bearing potential must agree to comply with any applicable contraceptive requirements of the protocol. If male, must agree to use an acceptable method of birth control, as defined in the protocol, during the study treatment administration period and for 90 days afterward if treated with maribavir, ganciclovir, valganciclovir, or cidofovir and for 180 days afterward if treated with foscarnet.
10. The participant must be able to swallow tablets, or receive tablets crushed and/or dispensed in water via nasogastric or orogastric tube.
11. The participant must be willing and have an understanding and ability to fully comply with study procedures and restrictions defined in the protocol.
12. The participant must be willing to provide necessary samples (example [e.g,] biopsy) for the diagnosis of tissue invasive CMV disease at baseline as determined by the Investigator.
13. The participant must have a life expectancy of >= 8 weeks.

Exclusion Criteria:

1. Have a current CMV infection that is considered refractory or resistant due to inadequate adherence to prior anti-CMV treatment, to the best knowledge of the Investigator.
2. Require ganciclovir, valganciclovir, foscarnet, or cidofovir administration for conditions other than CMV when study treatment is initiated (example: herpes simplex virus (HSV) coinfection requiring use of any of these agents after the randomization) or would need a coadministration with maribavir for CMV infection. NOTE: A participant who is not continuing with the same anti-CMV drug(s) (ganciclovir, valganciclovir or foscarnet) for the study treatment (if randomized to the investigator assigned anti-CMV treatment arm), must discontinue their use before the first dose of study drug. If participant is currently being treated with cidofovir and is assigned another anti-CMV therapy by the investigator, the participant must discontinue its use at least 14 days prior to randomization at Visit 2/Day 0 and the first dose of study treatment.
3. Be receiving leflunomide, letermovir, or artesunate when study treatment is initiated. NOTE: Participants receiving leflunomide must discontinue the use at least 14 days prior to randomization at Visit 2/Day 0 and the first dose of study treatment. Participants receiving letermovir must discontinue use at least 3 days prior to the first dose of study treatment. Participants receiving artesunate must discontinue the use prior to the first dose of study treatment.
4. Have severe vomiting, diarrhea, or other severe gastrointestinal illness within 24 hours prior to the first dose of study treatment that would preclude administration of oral/enteral medication.
5. Have known hypersensitivity to the active substance or to an excipient for a study treatment.
6. Have tissue invasive CMV disease with central nervous system involvement including the retina (example, CMV retinitis).
7. Have serum aspartate aminotransferase (AST) > 5 times upper limit of normal (ULN) at screening, or serum alanine aminotransferase (ALT) > 5 times ULN at screening, or total bilirubin >= 3.0 x ULN at screening (except for documented Gilbert's syndrome), by local or central lab. Participants with biopsy confirmed CMV hepatitis will not be excluded from study participation despite AST or ALT > 5 times ULN at screening.
8. Have known positive results for human immunodeficiency virus (HIV). Participants must have a confirmed negative HIV test result within 3 months of study entry or, if unavailable, be tested by a local laboratory during the screening period.
9. Require mechanical ventilation or vasopressors for hemodynamic support at the time of enrollment.
10. Be female and pregnant or breast feeding.
11. Have previously received maribavir.
12. Have received any investigational agent with known anti-CMV activity within 30 days before initiation of study treatment or investigational CMV vaccine at any time.
13. Have received any unapproved agent or device within 30 days before initiation of study treatment.
14. Have active malignancy with the exception of nonmelanoma skin cancer. Participants who have had a hematopoietic stem cell transplant (HSCT) and who experience relapse or progression of the malignancy as per investigator's opinion are not to be enrolled.
15. Be undergoing treatment for acute or chronic hepatitis C.
16. Have any clinically significant medical or surgical condition that, in the investigator's opinion, could interfere with the interpretation of study results, contraindicate the administration of the assigned study treatment, or compromise the safety or well-being of the participant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (134):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - AdventHealth, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Feinberg School of Medicine Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Chicago Medical Center, Maywood, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Weill-Cornell, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Health Sciences Center - PPDS, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Washington
  - Princess Alexandra Hospital, Brisbane
- Austria (2):
  - Tiroler Landeskrankenanstalten GmbH, Innsbruck
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Belgium (8):
  - UZ Antwerpen, Edegem, Antwerpen
  - Institut Jules Bordet, Brussels, Brussels Capital
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - AZ Sint-Jan AV, Bruges, West-Vlaanderen
  - ZNA Stuivenberg, Antwerp
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- University Hospital Center Zagreb, Zagreb, Croatia
- Copenhagen University Hospital, København Ø, Capital, Denmark
- France (23):
  - CHRU Brest - Hospital Cavale Blanche, Brest, Finistère
  - Hôpital de Rangueil, Toulouse, Haute-Garonne
  - Hopital Foch, Suresnes, Hauts-de-Seine
  - CHRU Rennes, Rennes, Ille-et-Vilaine
  - CHRU Bretonneau, Tours, Indre-et-Loire
  - CHRU Nantes, Nantes, Loire-Atlantique
  - Hôpital de La Croix Rousse, Lyon, Rhône
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Hopital Henri Mondor, Créteil, Val-de-Marne
  - Hôpital Paul Brousse, Villejuif, Val-de-Marne
  - CHU Amiens Hôpital Sud, Amiens
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU de GRENOBLE, Grenoble
  - CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - Groupement Hospitalier Edouard Herriot, Lyon
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - CHRU de Poitiers La Miletrie, Poitiers
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Hopital de Hautepierre, Strasbourg
  - Hôpital Civil, Strasbourg
- Germany (9):
  - University Clinic Heidelberg - PPDS, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Erlangen, Erlangen
  - University Clinic Heidelberg - PPDS, Heidelberg
  - LMU Klinikum der Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
- Italy (7):
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona, The Marches
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Singapore General Hospital (SGH), Singapore, Singapore
- Spain (10):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Cruces, Barakaldo
  - Fundacio Puigvert, Barcelona
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Centre Hospitalier Universitaire Vaudois, Lausanne, Vaud (fr), Switzerland
- United Kingdom (11):
  - University Hospital Coventry, Coventry, Birmingham
  - Birmingham Heartlands Hospital, West Midlands, Birmingham
  - Beatson West of Scotland Cancer Centre - PPDS, Glasgow, Glasgow City
  - Imperial College Healthcare NHS Trust, London, London, City of
  - Wythenshawe Hospital - PPDS, Wythenshawe, Manchester
  - Sheffield Childrens Hospital, Sheffield, Yorkshire
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - Royal Free Hospital, London
  - Manchester Royal Infirmary - PPDS, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rajagopalan K, Bullano M, Gelone D, Bo T, Taduka V, Syed SS. Real-world effectiveness and tolerability of post solid organ transplant patients with CMV switching from valganciclovir treatment to maribavir: analysis using lab-linked claims data in the United States. Expert Rev Anti Infect Ther. 2025 Aug;23(8):653-662. doi: 10.1080/14787210.2025.2517344. Epub 2025 Jun 27. PMID 40478680
- [Derived] Blumberg EA, Witzke O, Harber M, Ison MG, Saliba F, Kamar N, Sundberg AK, Gu J, Kumar D, La Hoz RM. Maribavir for refractory cytomegalovirus infection (with or without resistance) in solid organ transplant recipients: Subgroup analysis of the phase 3 randomized SOLSTICE study. J Heart Lung Transplant. 2025 Jun;44(6):986-994. doi: 10.1016/j.healun.2024.11.026. Epub 2024 Nov 28. PMID 39613120
- [Derived] Sun K, Fournier M, Sundberg AK, Song IH. Maribavir: Mechanism of action, clinical, and translational science. Clin Transl Sci. 2024 Jan;17(1):e13696. doi: 10.1111/cts.13696. PMID 38071422
- [Derived] Chou S, Alain S, Cervera C, Chemaly RF, Kotton CN, Lundgren J, Papanicolaou GA, Pereira MR, Wu JJ, Murray RA, Buss NE, Fournier M. Drug Resistance Assessed in a Phase 3 Clinical Trial of Maribavir Therapy for Refractory or Resistant Cytomegalovirus Infection in Transplant Recipients. J Infect Dis. 2024 Feb 14;229(2):413-421. doi: 10.1093/infdis/jiad293. PMID 37506264
- [Derived] Avery RK, Alain S, Alexander BD, Blumberg EA, Chemaly RF, Cordonnier C, Duarte RF, Florescu DF, Kamar N, Kumar D, Maertens J, Marty FM, Papanicolaou GA, Silveira FP, Witzke O, Wu J, Sundberg AK, Fournier M; SOLSTICE Trial Investigators. Maribavir for Refractory Cytomegalovirus Infections With or Without Resistance Post-Transplant: Results From a Phase 3 Randomized Clinical Trial. Clin Infect Dis. 2022 Sep 10;75(4):690-701. doi: 10.1093/cid/ciab988. PMID 34864943
- [Derived] Del Pozo Martin Y. 47th Annual Meeting of the EBMT. Lancet Haematol. 2021 May;8(5):e317-e318. doi: 10.1016/S2352-3026(21)00104-6. Epub 2021 Mar 31. No abstract available. PMID 33811823
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd74db2bf003ab46f3d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 94 sites in North America, Europe, and Asia Pacific between 22 December 2016 (first participant first visit) and 17 August 2020 (last participant last visit).
Pre-assignment Details: Participants with cytomegalovirus (CMV) infections were enrolled and randomized into two treatment groups: IAT (control), and Maribavir 400 mg. Participants randomized to IAT treatment arm, if met the stringent criteria for lack of improvement/worsening of CMV infection, considered eligible for entry into Maribavir rescue arm at Week 3 based on medical monitor review. As planned, combined data has been reported for IAT control group.
Groups:
- Investigator-assigned Anti-CMV Treatment (IAT): Participants received 1 or 2 of the 4 anti-CMV agents from the following: ganciclovir, valganciclovir, foscarnet, or cidofovir based on the investigator's discretion for the 8 week treatment period.
- Maribavir 400 mg: Participants received maribavir 400 milligram (mg) (2*200 mg tablets), orally, twice daily for the 8 week treatment period.
- Maribavir Rescue Arm: Participants with clear evidence of virologic failure (not just intolerance) after a minimum of 3 weeks of therapy with IAT entered maribavir rescue arm and received maribavir 400 mg (2*200 mg tablets), orally, twice daily for the 8 week treatment period.
Period: Period 1: Treatment Phase
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg | Maribavir Rescue Arm
Started | 117 | 235 | 0
Treated Participants | 116 | 234 | 0
IAT (Ganciclovir/ Valganciclovir) | 56 | 0 | 0
IAT (Foscarnet) | 47 | 0 | 0
IAT (Cidofovir) | 6 | 0 | 0
IAT (Foscarnet + Valganciclovir/Ganciclovir) | 7 | 0 | 0
Completed | 58 | 199 | 0
Not Completed | 59 | 36 | 0
Not completed — Investigator discretion | 1 | 1 | 0
Not completed — Adverse Event | 5 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Death | 8 | 24 | 0
Not completed — Withdrawal by Subject | 16 | 8 | 0
Not completed — Protocol Violation | 6 | 0 | 0
Not completed — Participants transitioned into maribavir rescue arm | 22 | 0 | 0
Period: Period 2: Maribavir Rescue Therapy
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg | Maribavir Rescue Arm
Started | 0 | 0 | 22
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 2
Not completed — Sponsor decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The randomized set consisted of all participants who had signed an informed consent and had begun some study procedures, and randomized to the study.
Groups:
- Maribavir 400 mg: Participants received maribavir 400 mg (2*200 mg tablets), orally, twice daily for the 8 week treatment period.
- Total: Total of all reporting groups
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg | Total
Number analyzed (Participants) | 117 | 235 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.80) | 53.8 (13.39) | 53.0 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 87 | 139
  Male | 65 | 148 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 21
  Not Hispanic or Latino | 95 | 198 | 293
  Unknown or Not Reported | 15 | 23 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 9 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 29 | 47
  White | 87 | 179 | 266
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 18 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Confirmed Clearance of Plasma Cytomegalovirus (CMV) Deoxyribonucleic Acid (DNA) (CMV Viremia Clearance) at End of Week 8
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration less than (<) lower limit of quantification (LLOQ) that is, <137 International Units per milliliter (IU/mL) when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive postbaseline samples, separated by at least 5 days. Percentage of participants with confirmed CMV viremia clearance at end of study Week 8 regardless of whether either study-assigned treatment was discontinued before the end of the stipulated 8 weeks of therapy, and could not have received alternative anti-CMV treatment were reported.
Time Frame: Week 8
Population: The randomized set consisted of all participants who had signed informed consent and had begun some study procedures and were randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 23.9 | 55.7
Statistical Analysis 1: Comparison: Investigator-assigned Anti-CMV Treatment (IAT) vs Maribavir 400 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage of responders = 32.8, 95% CI 2-sided [22.80 to 42.74]

2. Secondary Outcome: Percentage of Participants Who Achieved Confirmed CMV Viremia Clearance and CMV Infection Symptom Control at End of Week 8, Followed by Maintenance of Treatment Effect at Week 16
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration <LLOQ that is, <137 IU/mL when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive postbaseline samples, separated by at least 5 days. CMV infection symptom control was defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline, or maintaining no symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline. Percentage of participants who achieved CMV viremia clearance and CMV infection symptom control at end of Week 8 through Week 16 were reported.
Time Frame: Up to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 10.3 | 18.7
Statistical Analysis 1: Comparison: Investigator-assigned Anti-CMV Treatment (IAT) vs Maribavir 400 mg; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel; Difference in percentage of responders = 9.5, 95% CI 2-sided [2.02 to 16.88]

3. Secondary Outcome: Percentage of Participants Who Achieved Confirmed CMV Viremia Clearance After Receiving 8 Weeks of Study-assigned Treatment
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration <LLOQ that is, <137IU/mL when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive postbaseline samples, separated by at least 5 days. Percentage of participants who achieved confirmed CMV viremia clearance after receiving 8 weeks study-assigned treatment at end of Week 8, and maintained this effect through 12, 16 and 20 were reported.
Time Frame: At Week 8 through Weeks 12, 16 and 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants
  At Week 8 | 18.8 | 54.9
  At Week 12 | 5.1 | 22.6
  At Week 16 | 5.1 | 18.7
  At Week 20 | 4.3 | 18.3

4. Secondary Outcome: Percentage of Participants Who Achieved Confirmed CMV Viremia Clearance and CMV Infection Symptom Control After Receiving 8 Weeks of Study-assigned Treatment Through Weeks 12, 16 and 20
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration <LLOQ that is, <137IU/mL when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive postbaseline samples, separated by at least 5 days. CMV infection symptom control was defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline, or maintaining no symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline. Percentage of participants who achieved confirmed CMV viremia clearance and CMV infection control after receiving 8 weeks study-assigned treatment at end of Week 8, and maintained this effect through 12, 16 and 20 were reported.
Time Frame: At Week 8 through Weeks 12, 16 and 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants
  At Week 8 | 18.8 | 54.9
  At Week 12 | 5.1 | 22.6
  At Week 16 | 5.1 | 18.7
  At Week 20 | 4.3 | 18.3

5. Secondary Outcome: Percentage of Participants Who Maintained CMV Viremia Clearance and CMV Infection Symptom Control at the End of Study Week 8 Through Weeks 12 and 20 Regardless of Whether Either Study-assigned Treatment Was Discontinued Before 8 Weeks of Therapy
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration <LLOQ that is, <137IU/mL when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive postbaseline samples, separated by at least 5 days. CMV infection symptom control was defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline or maintaining no symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline. Percentage of participants who maintained CMV viremia clearance and CMV infection symptom control at the end of study Week 8 through Weeks 12 and 20 regardless of whether either study-assigned treatment was discontinued before 8 weeks of therapy were reported.
Time Frame: At Week 8 through Weeks 12 and 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants
  At Week 8 | 23.9 | 55.7
  At Week 12 | 10.3 | 22.6
  At Week 20 | 9.4 | 18.3

6. Secondary Outcome: Percentage of Participants With Recurrence of CMV Viremia During the First 8 Weeks of Study Regardless of Whether Study-assigned Treatment Was Discontinued Before 8 Weeks of Therapy
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration greater than or equal to (>=) LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance, regardless of whether either study-assigned treatment was discontinued before the end of the stipulated 8 weeks of therapy. Percentage of participants with recurrence of CMV viremia during the first 8 weeks of study regardless of whether study-assigned treatment was discontinued before 8 weeks of therapy were reported.
Time Frame: At Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 12.3 | 17.9

7. Secondary Outcome: Percentage of Participants With Recurrence of CMV Viremia During the 12 Weeks Follow-up Period Regardless of Whether Study-assigned Treatment Was Discontinued Before 8 Weeks of Therapy
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance, regardless of whether either study-assigned treatment was discontinued before the end of the stipulated 8 weeks of therapy. Percentage of participants with recurrence of CMV viremia during the 12 weeks follow-up period regardless of whether study-assigned treatment was discontinued before 8 weeks of therapy were reported.
Time Frame: End of Week 8 up to Week 20 (12 weeks follow-up period)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 21.5 | 38.6

8. Secondary Outcome: Percentage of Participants With Recurrence of CMV Viremia at Any Time on Study Regardless of Whether Study-assigned Treatment Was Discontinued Before 8 Weeks of Therapy
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance, regardless of whether either study-assigned treatment was discontinued before the end of the stipulated 8 weeks of therapy. Percentage of participants with recurrence of CMV viremia during at any time on study regardless of whether study-assigned treatment was discontinued before 8 weeks of therapy were reported.
Time Frame: Baseline up to Week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 33.8 | 56.5

9. Secondary Outcome: Percentage of Participants Who Completed 8 Weeks of Study-assigned Treatment With Recurrence of CMV Viremia During the First 8 Weeks of the Treatment
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants with recurrence of CMV viremia during the first 8 Weeks of the treatment who completed 8 weeks of study-assigned treatment were reported.
Time Frame: Baseline up to Week 8
Population: The randomized set consisted of all participants who had signed informed consent and had begun some study procedures and were randomized to the study. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 37 | 183
percentage of participants | 9.7 | 15.2

10. Secondary Outcome: Percentage of Participants Who Completed 8 Weeks of Study-assigned Treatment With Recurrence of CMV Viremia During the 12 Weeks of Follow-up Period
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants who completed 8 weeks of study-assigned treatment with recurrence of CMV viremia during the 12 weeks of follow-up period were reported.
Time Frame: End of Week 8 up to Week 20 (12 weeks follow-up period)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 37 | 183
percentage of participants | 35.5 | 40.9

11. Secondary Outcome: Percentage of Participants Who Completed 8 Weeks of Study-assigned Treatment With Recurrence of CMV Viremia During the 20 Weeks of Study
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants with Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants who completed 8 weeks of study-assigned treatment with recurrence of CMV viremia during the 20 weeks of study were reported.
Time Frame: Baseline up to Week 20
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 37 | 183
percentage of participants | 45.2 | 56.1

12. Secondary Outcome: Percentage of Participants With Recurrence of CMV Viremia While on Study-assigned Treatment
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants with recurrence of CMV viremia while on study-assigned treatment period were reported.
Time Frame: Baseline up to termination of study treatment (up to Week 8)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 4.6 | 15.8

13. Secondary Outcome: Percentage of Participants With Recurrence of CMV Viremia While Off Study-assigned Treatment During Follow-up Period
Description: Recurrence of CMV viremia was defined as plasma CMV DNA concentration >=LLOQ when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants with recurrence of CMV viremia while off study-assigned treatment during follow-up period were reported.
Time Frame: Termination of study treatment (Week 8) up to the End of the Study (Week 20)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
percentage of participants | 29.2 | 40.8

14. Secondary Outcome: Number of Participants Who Had Maribavir CMV Resistance at Baseline
Description: Resistance-associated amino acid substitutions (RASs) to maribavir are known to generally map to the pUL97 and pUL27 genes. Genotyping was performed to identify RASs mapping to the pUL97 and pUL27 genes. Number of participants who had maribavir CMV resistance at baseline were reported.
Time Frame: At Baseline
Population: The combination of maribavir resistance set (MRS) and non-MRS set (MRS+non-MRS) included all participants in modified randomized set who had been randomized in the study and who had taken any dose of study-assigned treatment with evaluable CMV genotypic data at baseline with or without pre-existing known maribavir RASs in pUL97 and/or pUL27. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir Rescue Arm | Maribavir 400 mg
Number analyzed (Participants) | 100 | 17 | 214
Participants
  RASs associated with pUL97 only | 3 | 1 | 0
  RASs associated with pUL27 only | 0 | 0 | 1
  RASs associated with pUL97 and pUL27 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants Who Had Post-baseline Resistance to Maribavir
Description: Resistance-associated amino acid substitutions (RASs) to maribavir are known to generally map to the pUL97 and pUL27 genes. Genotyping was performed to identify RASs mapping to the pUL97 and pUL27 genes. Number of participants who had post-baseline resistance to maribavir were reported.
Time Frame: After first dose of study drug up to Week 20
Population: The combination of maribavir resistance set (MRS) and non-MRS set (MRS+non-MRS) included all participants in modified randomized set who had been randomized in the study and who had taken any dose of study-assigned treatment with evaluable CMV genotypic data at baseline with or without pre-existing known maribavir RASs in pUL97 and/or pUL27.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir Rescue Arm | Maribavir 400 mg
Number analyzed (Participants) | 100 | 17 | 214
Participants
  RASs associated with pUL97 only | 0 | 4 | 45
  RASs associated with pUL27 only | 0 | 0 | 0
  RASs associated with pUL97 and pUL27 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With All-cause Mortality by the End of the Study
Description: All-cause mortality was analyzed by the end of study regardless of the use of rescue treatment or alternative anti-CMV treatment. Number of participants who died during the entire study period were reported.
Time Frame: From enrollment up to end of study (approximately 44 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
Participants | 13 | 27

17. Secondary Outcome: Time to All Cause Mortality
Description: The time to all-cause mortality by the end of the study participation in days was calculated. Participants who were alive at the last study follow-up (regardless of use of rescue or alternative anti-CMV treatment), withdrew from study or were lost to follow-up were censored at the date of last contact.
Time Frame: From enrollment to last serious adverse event (SAE) follow-up (approximately Week 28)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir 400 mg
Number analyzed (Participants) | 117 | 235
days | 73.0 [13.0 to 186.0] | 55.0 [3.0 to 182.0]
Statistical Analysis 1: Comparison: Investigator-assigned Anti-CMV Treatment (IAT) vs Maribavir 400 mg; Test type: Other; p = 0.647, Log Rank; Two-sided p-value comparing treatment groups was calculated from the log rank test by Kaplan-Meier Method; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.549 to 2.357] — Stratified Cox regression model was used as transplant type and baseline plasma CMV DNA level as stratification factors

18. Secondary Outcome: Percentage of Participants Who Achieved Confirmed Clearance of Plasma CMV DNA (CMV Viremia Clearance) at End of Week 8 After Starting Maribavir Rescue Treatment
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration <LLOQ that is, <137 IU/mL when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV Test in 2 consecutive postbaseline samples, separated by at least 5 days, regardless of whether the rescue treatment was discontinued before the end of the stipulated 8 weeks of therapy. Percentage of participants who achieved confirmed CMV viremia clearance at end of Week 8 after starting maribavir rescue treatment were reported.
Time Frame: From start of maribavir rescue treatment through 8 weeks
Population: The rescue set consisted of all participants who entered the rescue arm and received any dose of maribavir as rescue therapy. As planned, this OM was assessed only in maribavir rescue arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maribavir Rescue Arm
Number analyzed (Participants) | 22
percentage of participants | 50.0 [28.22 to 71.78]

19. Secondary Outcome: Percentage of Participants Receiving Maribavir Rescue Treatment Who Achieved Confirmed CMV Viremia Clearance and CMV Infection Symptom Control at Week 8 With Maintenance of Effect Through Week 16
Description: Confirmed CMV viremia clearance was defined as plasma CMV DNA concentration <LLOQ that is, <137 IU/mL when assessed by COBAS® AmpliPrep/COBAS® TaqMan® CMV test in 2 consecutive postbaseline samples, separated by at least 5 days. CMV infection symptom control was defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline, or maintaining no symptoms of tissue invasive CMV disease or CMV syndrome for participants asymptomatic at baseline. Percentage of participants receiving maribavir rescue treatment who achieved confirmed CMV viremia clearance and CMV infection symptom control at Week 8 with maintenance of effect through Week 16 were reported.
Time Frame: Up to Week 16
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maribavir Rescue Arm
Number analyzed (Participants) | 22
percentage of participants | 27.3 [10.73 to 50.22]

20. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs During the On-treatment Observation Period
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Serious AE was any untoward medical occurrence (whether considered to be related to study-assigned treatment or not) that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital abnormality/birth defect, or was an important medical event. TEAEs was defined as any adverse events (classified by preferred term) that had a start date on or after the first dose of study treatment or that had a start date before the date of first dose of study treatment, but increased in severity after the first dose of study treatment.
Time Frame: Baseline up to 7 days or 21 days (if cidofovir used) after the last dose of study treatment (up to Week 8)
Population: The safety set consisted of all participants who had taken any dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Investigator-assigned Anti-CMV Treatment (IAT): Participants received 1 or 2 of the 4 anti-CMV agents from the following: ganciclovir, valganciclovir, foscarnet, or cidofovir based on the investigator's discretion Participants received 1 or 2 of the 4 anti-CMV agents from the following: ganciclovir, valganciclovir, foscarnet, or cidofovir based on the investigator's discretion for the 8 week treatment period.
Arm/Group | Investigator-assigned Anti-CMV Treatment (IAT) | Maribavir Rescue Arm | Maribavir 400 mg
Number analyzed (Participants) | 116 | 22 | 234
Participants
  TEAEs | 106 | 22 | 228
  Serious TEAEs | 43 | 11 | 90

21. Secondary Outcome: Predose Concentration (Cmin) of Maribavir
Description: Cmin of maribavir was reported.
Time Frame: Predose at Week 1, 4 and 8
Population: The pharmacokinetic set consisted of all participants who had taken any dose of study treatment and who had plasma samples drawn and tested for maribavir concentrations. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure and "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Maribavir 400 mg | Maribavir Rescue Arm
Number analyzed (Participants) | 208 | 20
micrograms per milliliter (mcg/mL)
  Cmin at Week 1 | 8.77 (7.88) | 8.57 (6.28)
  Cmin at Week 4: number analyzed (Participants) | 177 | 16
  Cmin at Week 4 | 7.59 (7.05) | 5.75 (3.99)
  Cmin at Week 8: number analyzed (Participants) | 168 | 18
  Cmin at Week 8 | 7.19 (6.41) | 5.65 (4.47)

22. Secondary Outcome: Area Under the Concentration Time Curve Over the 12-hour Dosing Interval at Steady State (AUC0-tau) of Marivabir for Adolescent Participants
Description: AUC0-tau of maribavir for adolescent participants was planned to be reported.
Time Frame: Week 1: Pre-morning dose and 1, 2, 3, 4, 6, 8 and 12 hours post morning dose, Week 4: Pre-morning dose, and Week 8: Pre-morning dose and 2-4 hour post morning dose
Population: The pharmacokinetic set consisted of all participants who had taken any dose of study treatment and who had plasma samples drawn and tested for maribavir concentrations. This OM was planned to be analyzed only in adolescent participants. Data was not collected and analyzed as adolescent participants were not enrolled in this study. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Arm/Group | Maribavir 400 mg | Maribavir Rescue Arm
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Maribavir for Adolescent Participants
Description: Cmax of maribavir for adolescent participants was planned to be reported.
Time Frame: Week 1: Pre-morning dose and 1, 2, 3, 4, 6, 8 and 12 hours post morning dose
Population: as for outcome 22
Arm/Group | Maribavir 400 mg | Maribavir Rescue Arm
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Time When Maximum Concentration is Observed (Tmax) of Maribavir for Adolescent Participants
Description: Tmax of maribavir for adolescent participants was planned to be reported.
Time Frame: Week 1: Pre-morning dose and 1, 2, 3, 4, 6, 8 and 12 hours post morning dose
Population: as for outcome 22
Arm/Group | Maribavir 400 mg | Maribavir Rescue Arm
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Apparent Oral Clearance (CL/F) of Maribavir for Adolescent Participants
Description: Apparent oral clearance (CL/F) of maribavir for adolescent participants was planned to be reported.
Time Frame: Week 1: Pre-morning dose and 1, 2, 3, 4, 6, 8 and 12 hours post morning dose
Population: as for outcome 22
Arm/Group | Maribavir 400 mg | Maribavir Rescue Arm
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Maribavir for Adolescent Participants
Description: Apparent volume of distribution (Vz/F) of maribavir for adolescent participants was planned to be reported.
Time Frame: Week 1: Pre-morning dose and 1, 2, 3, 4, 6, 8 and 12 hours post morning dose
Population: as for outcome 22
Arm/Group | Maribavir 400 mg | Maribavir Rescue Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (approximately 44 months)
Groups:
- IAT: Ganciclovir/ Valganciclovir: Participants received ganciclovir intravenously or valganciclovir orally based on the the investigator's discretion for the 8 week treatment period.
- IAT: Foscarnet: Participants received foscarnet intravenously based on investigator's discretion for the 8 week treatment period.
- IAT: Cidofovir: Participants received cidofovir intravenously based on the investigator's discretion for the 8 week treatment period.
- IAT: Foscarnet + Ganciclovir/ Valganciclovir: Participants received foscarnet intravenously in combination with ganciclovir intravenously or valganciclovir orally based on investigator's discretion for the 8 week treatment period.
Arm/Group | IAT: Ganciclovir/ Valganciclovir | IAT: Foscarnet | IAT: Cidofovir | IAT: Foscarnet + Ganciclovir/ Valganciclovir | Maribavir 400 mg | Maribavir Rescue Arm
All-Cause Mortality (participants affected / at risk) | 6/56 | 7/47 | 0/6 | 0/7 | 27/234 | 0/22
Serious Adverse Events (participants affected / at risk) | 33/56 | 26/47 | 3/6 | 1/7 | 131/234 | 14/22
Other Adverse Events (participants affected / at risk) | 54/56 | 43/47 | 5/6 | 7/7 | 229/234 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IAT: Ganciclovir/ Valganciclovir (N=56) | IAT: Foscarnet (N=47) | IAT: Cidofovir (N=6) | IAT: Foscarnet + Ganciclovir/ Valganciclovir (N=7) | Maribavir 400 mg (N=234) | Maribavir Rescue Arm (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug interaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Treatment failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Cytomegalovirus mucocutaneous ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis cytomegalovirus (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 1 (1)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral load increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 13 (14) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal transplant failure (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus enterocolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IAT: Ganciclovir/ Valganciclovir (N=56) | IAT: Foscarnet (N=47) | IAT: Cidofovir (N=6) | IAT: Foscarnet + Ganciclovir/ Valganciclovir (N=7) | Maribavir 400 mg (N=234) | Maribavir Rescue Arm (N=22)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 10 (12) | 1 (2) | 1 (1) | 31 (36) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 2 (2) | 0 (0) | 1 (1) | 12 (15) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 19 (41) | 8 (17) | 0 (0) | 1 (2) | 38 (92) | 7 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 18 (19) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 22 (26) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8) | 1 (1) | 0 (0) | 1 (1) | 9 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7) | 2 (3) | 0 (0) | 1 (2) | 14 (14) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 10 (15) | 1 (2) | 1 (4) | 67 (92) | 10 (13)
Nausea (Gastrointestinal disorders) | 12 (17) | 16 (19) | 2 (2) | 2 (4) | 67 (88) | 5 (6)
Vomiting (Gastrointestinal disorders) | 13 (16) | 9 (10) | 1 (1) | 2 (2) | 46 (69) | 2 (3)
Fatigue (General disorders) | 10 (10) | 5 (5) | 0 (0) | 1 (1) | 36 (38) | 3 (3)
Oedema peripheral (General disorders) | 5 (7) | 7 (10) | 0 (0) | 2 (2) | 26 (27) | 3 (3)
Pyrexia (General disorders) | 12 (15) | 10 (11) | 2 (2) | 0 (0) | 32 (48) | 5 (6)
Cytomegalovirus viraemia (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 2 (2) | 32 (33) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 18 (19) | 1 (1)
Immunosuppressant drug level increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 21 (23) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 1 (1) | 1 (1) | 23 (25) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 8 (12) | 0 (0) | 1 (1) | 13 (16) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (7) | 9 (10) | 1 (1) | 0 (0) | 14 (17) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 16 (17) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 2 (2) | 1 (1) | 2 (3) | 20 (23) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 88 (95) | 1 (1)
Headache (Nervous system disorders) | 9 (11) | 9 (10) | 0 (0) | 3 (3) | 30 (34) | 2 (3)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 21 (21) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 7 (9) | 0 (0) | 0 (0) | 26 (33) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 1 (1) | 1 (1) | 22 (28) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 23 (24) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 6 (7) | 0 (0) | 1 (1) | 15 (15) | 1 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 10 (11) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BK virus infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 7 (8) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 25 (30) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 13 (16) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 12 (13) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 4 (5) | 1 (4) | 0 (0) | 0 (0) | 5 (6) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 6 (10) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 11 (13) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 7 (9) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 17 (20) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 8 (9) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 13 (15) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 12 (16) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (10) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 12 (12) | 0 (0)
Systemic bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 8 (12) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 10 (11) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 17 (22) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 7 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02931539/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02931539/SAP_001.pdf